CLINICAL TRIAL: NCT00001753
Title: Study of Temperature Effects on Skeletal Muscle Aerobic Energy Metabolism
Brief Title: Study of the Effects of Temperature on Metabolism in Human Muscle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980166; 98-H-0166
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Healthy
Keywords: Exercise; MRI; MRS; Normal Volunteer; Tibialix Anterior
MeSH Terms: conditions — Motor Activity | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: Magnetic resonance imaging

SUMMARY:
This study will examine the role of temperature in changing energy metabolism in human muscle. In order to do this, researchers will use magnetic resonance imaging (MRI) to provide information about how parts of muscle operate during exercise.

Magnetic resonance imaging (MRI) is a diagnostic tool that creates high quality images of the human body without the use of X-ray (radiation). In this study, MRI will be used to measure the temperature and energy level of specific muscles during rest and exercise. In addition, the muscles being tested will be heated and cooled to see if temperature directly affects levels of energy in muscle.

DETAILED DESCRIPTION:
This study will examine the role of temperature in modulating aspects of energy metabolism in human skeletal muscle. Tests will be conducted at rest and during concentric dorsiflexion exercise of the Tibialis anterior (TA) muscle using an existing custom-designed dynamometer in conjunction with mild local heating and cooling. Magnetic resonance spectroscopy (MRS), performed in a 4-tesla whole-body NMR system, will be used to non-invasively measure muscle temperature and energy-state. Specifically these tests will assess the extent to which temperature changes occur during aerobic exercise and how small temperature changes affect mitochondrial function in-vivo.

ELIGIBILITY:
Ages 18 to 50.

Male and female subjects.

Capable of giving informed consent.

Healthy normal volunteers.

No cardiac pacemaker of implantable defibrillator.

No aneurysm clip.

No neural stimulator (e.g. TENS-unit).

No ear implant of any type.

No metal in the eye (e.g. from machining).

No implanted device (e.g. insulin pump, drug infusion device).

No metallic foreign body, shrapnel, or bullet.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17
Dates: Start 1998-09; Study Completion 2000-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fowler MD, Ryschon TW, Wysong RE, Combs CA, Balaban RS. Normalized metabolic stress for 31P-MR spectroscopy studies of human skeletal muscle: MVC vs. muscle volume. J Appl Physiol (1985). 1997 Sep;83(3):875-83. doi: 10.1152/jappl.1997.83.3.875. PMID 9292476